CLINICAL TRIAL: NCT06627764
Title: SER Familia: A Family-Based Intervention Addressing Syndemic Conditions Among Latino Immigrant Families
Acronym: SER Familia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: Pro00114672; 1R01MD018920-01A1 (NIH)
Record Dates: First submitted 2024-10-03; First posted 2024-10-04 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-02

CONDITIONS: Substance Abuse; Intimate Partner Violence (IPV); HIV Infections; Depression; Anxiety
Keywords: Family; Stress; Resilience
MeSH Terms: conditions — Substance-Related Disorders; HIV Infections; Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Familia SER (Salud, Estrés y Resilencia) Group (Experimental): Participants will attend six intervention sessions.
  Interventions: Behavioral: SER Familia
- Control Group (No Intervention): Participants will not receive SER Familia sessions.

INTERVENTIONS:
Behavioral: SER Familia — SER Familia is a six-session intervention co-developed and delivered by community health workers (CHWs) that uses strategies to reduce acculturative stress, promote resilience, improve parent-child and family level health, while simultaneously helping families maintain strong social networks and better navigate community resources to address social determinants of health (SDOH).
  Arms: Familia SER (Salud, Estrés y Resilencia) Group

SUMMARY:
This study aims to prevent syndemic health conditions by decreasing acculturative stress and promoting resilience via SER Familia (Salud, Estrés y Resilencia en Familias/ Health, Stress, and Resilience in Families), a family-based intervention. SER Familia is a six-session intervention co-developed and delivered by community health workers (CHWs) that uses strategies to reduce acculturative stress, promote resilience, improve parent-child and family level health, while simultaneously helping families maintain strong social networks and better navigate community resources to address social determinants of health (SDOH). More specifically, investigators aim to: 1) Examine the efficacy of SER Familia to prevent or reduce the syndemic comprised of substance abuse, IPV, HIV risk, depression, and anxiety among Parents and Youth; and 2) Identify how individual, family, and community mechanisms of change related to acculturative stress and resilience mediates the effect of SER Familia.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants must identify as Hispanic/Latino/a/x/e,
* be a first generation immigrant parent or parental figure (Parent)
* have a child (Youth) aged 12-17
* speak English and/or Spanish

Exclusion Criteria:

* Families planning to move within two years will be excluded

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in Parent Acculturative stress as measured by the Hispanic Stress Inventory (HSI-2) Immigrant Version | From Enrollment to end of treatment at 6 weeks
  The immigrant version of the HSI-2 includes 10 stress subscales. For each item, participants indicated whether they had experienced the stressor (Yes / No). If participants reported experiencing a stressor, then they rated how stressful the event was on a 5-point Likert scale (1= Not at all worried / tense; 2 = A little worried / tense; 3 = Moderately worried / tense; 4 = Very worried/ tense; 5 = Extremely worried/ tense). The total score ranges from 94 to 470, where a higher score indicates greater stress.
Change in Youth Acculturative stress as measured by the Hispanic Stress Inventory - Adolescent (HSI-A) | From Enrollment to end of treatment at 6 weeks
  The HSI-A includes 8 stress subscales. For each item, participants indicated whether they had experienced the stressor (Yes / No). If participants reported experiencing a stressor, then they rated how stressful the event was on a 5-point Likert scale (1= Not at all worried / tense; 2 = A little worried / tense; 3 = Moderately worried / tense; 4 = Very worried/ tense; 5 = Extremely worried/ tense). The total score ranges from 72 to 360, where a higher score indicates greater stress.
Change in individual resilience as measured by the 25-item Resiliency Scale | From Enrollment to end of treatment at 6 weeks
  The Resiliency Scale uses a 7-point Likert scale to assess how much a respondent agrees or disagrees with statements. The possible total score ranges from 25 to 175, with higher scores indicating greater resilience. Scores above 145 indicate high resilience, 121 to 145 indicate moderate resilience, and below 120 indicate low resilience.
Change in PROMIS (Patient-Reported Outcomes Measurement Information System) Global Health | From Enrollment to end of treatment at 6 weeks
  The PROMIS Global Health score ranges from 10 to 50, where a higher score indicates better overall health.

OTHER OUTCOMES:
Perceptions of the impact of SER Familia on Parents and Youth as measured by semi-structured interviews | From end of treatment at 6 weeks to the end of year two
  Exemplar questions include: 1) How did the program influence your resilience against family stress?; 2) What impact did the program have on your relationship with your parents/children?; 3) How did your parents/child's behaviors change throughout the program and after?; 4) How did those changes influence you and your family?; 5) What new connections or resources were you able to access during the program?; 6) What impact did this have on you, your family, or your community? 7) How did the impact of SER Familia influence the family over the past year (i.e., for 12-month follow-up)?

CONTACTS AND LOCATIONS:
Locations (1):
- Duke School of Nursing, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No